CLINICAL TRIAL: NCT01954108
Title: Hyaluronan in the Treatment of Painful Achilles Tendinopathy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TRB Chemedica AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OTENA-INT-2013-03; CIV-13-07-011543 (Other: EUDAMED)
Record Dates: First submitted 2013-09-26; First posted 2013-10-01 (Estimated); Last update posted 2015-11-09 (Estimated); Status verified 2015-11

CONDITIONS: Tendinopathy
Keywords: tendinopathy; hyaluronan; tendon; hyaluronic acid; extracorporeal shock wave
MeSH Terms: conditions — Tendinopathy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ESWT (Extracorporal Shock Wave Therapy) (Other): Three applications in weekly interval.
  Interventions: Device: ESWT
- hyaluronic acid sodium salt (Active Comparator): Two injections of 2% (40 milligrams (mg) / 2 millilitres (ml)) hyaluronan in weekly interval.
  Interventions: Device: hyaluronic acid sodium salt

INTERVENTIONS:
Device: hyaluronic acid sodium salt
  Other Names: OSTENIL® TENDON
  Arms: hyaluronic acid sodium salt
Device: ESWT
  Arms: ESWT (Extracorporal Shock Wave Therapy)

SUMMARY:
The primary objective of this study is to compare OSTENIL® TENDON (2% hyaluronan) and Extracorporeal Shock Wave (ESWT) therapy in the treatment of painful Achilles tendinopathy.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between 18 and 75 years of age.
* Good general health condition.
* Signed written informed consent.
* Painful Achilles midportion tendinopathy since more or equal than 6 weeks.
* Pain according to VAS (Huskisson, 100 mm) more or equal than 40 mm.
* Ensured compliance of subjects over the whole study period.

Exclusion Criteria:

* Concomitant or previous participation in a clinical investigation within the last 3 months prior to study inclusion.
* Infection or relevant skin disease at study relevant site.
* Blood coagulation disorder or intake of blood thinner (e.g. Marcumar).
* Known hypersensitivity to hyaluronic acid (HA) preparations or to the constituents mannitol, sodium chloride, disodium phosphate and sodium dihydrogenphosphate.
* Contra-indications for ESWT application in study relevant area (e.g. recent surgery, malignant tumour, local osteomyelitis or open epiphysis).
* Severe intercurrent illness (e.g. uncontrolled diabetes mellitus, peripheral neuropathy), which in the opinion of the investigator, may put the patient at risk when participating in the study, or affect the patient's ability to take part in the study.
* Concomitant disease at study relevant site (e.g. insertion tendinopathy at Achilles tendon) influencing study evaluation.
* Diseases or characteristics judged by the investigator to be incompatible with the assessments and/or procedures for the study evaluation.
* Intake of concomitant medications not allowed which might interfere with the functional assessment of the study (e.g. immunosuppressive drugs within the last 3 months).
* Previous therapies (except non-steroidal anti-inflammatory drugs (NSAID)) at study relevant site within the last 4 weeks prior to study inclusion.
* Use of NSAIDs within the last week prior to study treatment.
* Recent history of drug and/or alcohol abuse (within the last 6 months).
* Pregnant or lactating females.
* Participants of childbearing age (pre-menopausal) who do not accept the use of methods of birth control with pearl index of at least 1 (i.e. oral contraceptives, vaginal ring, hormone-releasing Intrauterine Device (IUD), implants, depot syringes, hormone patch, double barrier method, tubal ligation, vasectomised partner,…) during the treatment period and the first 4 weeks of follow-up period.
* Subjects not capable of contracting and of understanding the nature, risks, significance and implications of the clinical investigation and unable to form a rational intention in the light of these facts.
* Subjects unable to understand informed consent or having a high probability of non compliance to the study procedures and / or non completion of the study according to investigator's judgement (e.g. illiteracy, insufficient knowledge of local language).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2013-12; Primary Completion 2015-07 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Victorian Institute of Sports Assessment-Achilles (VISA-A score) | Day 90 (plus or minus 3 days)
  The validated questionnaire will be used to evaluate the outcome in Achilles tendinopathy. The score ranges from '0' to '100' whereas '0' denotes 'no activity / maximum pain' and '100' denote 'maximum activity / no pain'.

SECONDARY OUTCOMES:
Victorian Institute of Sports Assessment-Achilles (VISA-A score) | Day 0
  The validated questionnaire will be used to evaluate the outcome in Achilles tendinopathy. The score ranges from '0' to '100' whereas '0' denotes 'no activity / maximum pain' and '100' denote 'maximum activity / no pain'.
Victorian Institute of Sports Assessment-Achilles (VISA-A score) | Day 7 (plus or minus 1 day)
  The validated questionnaire will be used to evaluate the outcome in Achilles tendinopathy. The score ranges from '0' to '100' whereas '0' denotes 'no activity / maximum pain' and '100' denote 'maximum activity / no pain'.
Victorian Institute of Sports Assessment-Achilles (VISA-A score) | Day 28 (plus or minus 3 days)
  The validated questionnaire will be used to evaluate the outcome in Achilles tendinopathy. The score ranges from '0' to '100' whereas '0' denotes 'no activity / maximum pain' and '100' denote 'maximum activity / no pain'.
Victorian Institute of Sports Assessment-Achilles (VISA-A score) | Day 180 (plus or minus 3 days)
  The validated questionnaire will be used to evaluate the outcome in Achilles tendinopathy. The score ranges from '0' to '100' whereas '0' denotes 'no activity / maximum pain' and '100' denote 'maximum activity / no pain'.
Visual Analogue Scale of pain (VAS; 100 mm) | Day 0
  Intensity of pain will be evaluated on the Huskisson VAS pain scale on which 0 mm indicate 'no pain' and 100 mm indicate 'extreme pain'.
Visual Analogue Scale of pain (VAS; 100 mm) | Day 7 (plus or minus 1 day)
  Intensity of pain will be evaluated on the Huskisson VAS pain scale on which 0 mm indicate 'no pain' and 100 mm indicate 'extreme pain'.
Visual Analogue Scale of pain (VAS; 100 mm) | Day 28 (plus or minus 3 days)
  Intensity of pain will be evaluated on the Huskisson VAS pain scale on which 0 mm indicate 'no pain' and 100 mm indicate 'extreme pain'.
Visual Analogue Scale of pain (VAS; 100 mm) | Day 90 (plus or minus 3 days)
  Intensity of pain will be evaluated on the Huskisson VAS pain scale on which 0 mm indicate 'no pain' and 100 mm indicate 'extreme pain'.
Visual Analogue Scale of pain (VAS; 100 mm) | Day 180 (plus or minus 3 days)
  Intensity of pain will be evaluated on the Huskisson VAS pain scale on which 0 mm indicate 'no pain' and 100 mm indicate 'extreme pain'.
Patient's and investigator's global evaluation of study-relevant tendon complaints | Day 7 (plus or minus 1 day)
  Measured by Clinical Global Impression (CGI) 7-point scale, ranking from 'very much improved' to 'very much worse' condition.
Patient's and investigator's global evaluation of study-relevant tendon complaints | Day 28 (plus or minus 3 days)
  Measured by Clinical Global Impression (CGI) 7-point scale, ranking from 'very much improved' to 'very much worse' condition.
Patient's and investigator's global evaluation of study-relevant tendon complaints | Day 90 (plus or minus 3 days)
  Measured by Clinical Global Impression (CGI) 7-point scale, ranking from 'very much improved' to 'very much worse' condition.
Patient's and investigator's global evaluation of study-relevant tendon complaints | Day 180 (plus or minus 3 days)
  Measured by Clinical Global Impression (CGI) 7-point scale, ranking from 'very much improved' to 'very much worse' condition.
Clinical Parameters | Day 0
  * Redness
  * Warmth
  * Swelling
  * Tenderness on palpation
  * Crepitus on motion
  * Accumulation of tissue fluid
  Measured by 5-point scale, ranking from 'none' to 'extreme' intensity.
Clinical Parameters | Day 7 (plus or minus 1 day)
  * Redness
  * Warmth
  * Swelling
  * Tenderness on palpation
  * Crepitus on motion
  * Accumulation of tissue fluid
  Measured by 5-point scale, ranking from 'none' to 'extreme' intensity.
Clinical Parameters | Day 28 (plus or minus 3 days)
  * Redness
  * Warmth
  * Swelling
  * Tenderness on palpation
  * Crepitus on motion
  * Accumulation of tissue fluid
  Measured by 5-point scale, ranking from 'none' to 'extreme' intensity.
Clinical Parameters | Day 90 (plus or minus 3 days)
  * Redness
  * Warmth
  * Swelling
  * Tenderness on palpation
  * Crepitus on motion
  * Accumulation of tissue fluid
  Measured by 5-point scale, ranking from 'none' to 'extreme' intensity.
Clinical Parameters | Day 180 (plus or minus 3 days)
  * Redness
  * Warmth
  * Swelling
  * Tenderness on palpation
  * Crepitus on motion
  * Accumulation of tissue fluid
  Measured by 5-point scale, ranking from 'none' to 'extreme' intensity.
Frequency of test product-related Adverse Events | Up to Day 180

CONTACTS AND LOCATIONS:
Overall Officials: Thierry De Vroey, Dr. med., Principal Investigator — Universitair Ziekenhuis Antwerpen, Fysische Geneeskunde en Revalidatie; Nils Lynen, Dr. med., Principal Investigator — Praxiszentrum Orthopädie-Unfallchirurgie Nordrhein
Locations (2):
- Universitair Ziekenhuis Antwerpen, Fysische Geneeskunde en Revalidatie, Edegem, Belgium
- Praxiszentrum Orthopädie-Unfallchirurgie Nordrhein, Aachen, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Lynen N, De Vroey T, Spiegel I, Van Ongeval F, Hendrickx NJ, Stassijns G. Comparison of Peritendinous Hyaluronan Injections Versus Extracorporeal Shock Wave Therapy in the Treatment of Painful Achilles' Tendinopathy: A Randomized Clinical Efficacy and Safety Study. Arch Phys Med Rehabil. 2017 Jan;98(1):64-71. doi: 10.1016/j.apmr.2016.08.470. Epub 2016 Sep 14. PMID 27639439